CLINICAL TRIAL: NCT04047186
Title: Neoadjuvant Anti-PD-1 Therapy in Early Stage Non-small-cell Lung Cancer Presenting as Synchronous Ground-glass Nodules: a Pilot Study
Brief Title: Neoadjuvant Immunotherapy in Early Stage Non-small-cell Lung Cancer Presenting as Synchronous Ground-glass Nodules
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XiangNing Fu (Other)
Responsible Party: Sponsor-Investigator, XiangNing Fu, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019CR107
Record Dates: First submitted 2019-08-04; First posted 2019-08-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Multiple Pulmonary Nodules
Keywords: immunotherapy; Multiple Pulmonary Nodules; Lung Neoplasms
MeSH Terms: conditions — Multiple Pulmonary Nodules; Lung Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- neoadjuvant PD-1 group (Experimental): receiving neoadjuvant therapy of programmed death-1 (pd-1) immune checkpoint inhibitor
  Interventions: Drug: Tislelizumab Injection

INTERVENTIONS:
Drug: Tislelizumab Injection — Patients in the experimental group receive Tislelizumab Injection

SUMMARY:
Neoadjuvant Immunotherapy in Early Stage Non-small-cell Lung Cancer Presenting as Synchronous Ground-glass Nodules: a pilot study

DETAILED DESCRIPTION:
In many cases, non-small-cell lung cancer(NSCLC) manifested as synchronous ground-glass nodules(GGNs) and makes complete surgical resection impossible. At the same time, there is no good solution for the remaining GGNs after resection of the main lesion. Theoretically, pre-operative anti-PD-1 therapy is optimal for promoting anti-tumor immune response on the basis of maximum tumor mutational burden (TMB). In addition, neoadjuvant immunotherapy should have long-term anti-tumor effect even after surgery, because tumor recurrence may cause memory cells activation and differentiation. This is a pilot study to analysis the pathological remission rate of neoadjuvant immunotherapy and adverse events related to the treatment

ELIGIBILITY:
Inclusion Criteria:

* not less than two GGNs on chest CT
* at least one lesion is diagnosed as NSCLC from biopsy pathology
* no contraindication for surgery
* ECOG score of 0 or 1
* no detectable evidence of distant metastasis

Exclusion Criteria:

* medical history of malignancy
* pregnant or breeding period
* severe organ failure (heart, liver, kidney, and lung)
* high risk of cerebral-cardiovascular evens
* infection out of control
* received or receiving chemo- and radiotherapy
* history of severe reaction due to allergy or hypersensitivity
* severe mental disorder
* currently been enrolled in other trials
* autoimmune or chronic inflammatory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | twelve weeks

SECONDARY OUTCOMES:
treatment-related adverse events | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital Affiliated to Huazhong Technology Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
According to regulation of institution, IPD can not be shared.